CLINICAL TRIAL: NCT02572466
Title: Study of High Sensitive Troponin-I Level in End-stage Renal Disease Patients Receiving Hemodialysis
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Khajohn Tiranathanagul, Assistant Professor, Chulalongkorn University
Other Study IDs: 271/57
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: End-stage Renal Disease
Keywords: high-sensitive troponin-I; End-stage renal disease; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ESRD group: 1. Aged 18 years or older.
  2. was diagnosed as End-stage renal disease for more than one year.
  3. Attend hemodialysis 3 times a week consistently for more than 6 months.
  4. Hemodialysis with Kt/V > 1.2
  5. No urine output or is less than 500 ml per day.
  6. No symptoms of myocardial infarction Or were hospitalized with the similar diagnosis during the two weeks.
  Interventions: Other: Hemodialysis
- Control group: 1. Aged 18 years or older.
  2. without kidney disease (eGFR > 60 ml/min/1.73m2)

INTERVENTIONS:
Other: Hemodialysis — ESRD group received long-term hemodialysis
  Groups: ESRD group

SUMMARY:
This study objective is to compare the high sensitive troponin-I level in end-stage renal disease patients received hemodialysis without acute cardiovascular event with healthy population. The investigators also determine the effect of hemodialysis on troponin I level as the secondary objective.

DETAILED DESCRIPTION:
Human cardiac Troponin I (cTnI) is an composition of Troponin which is found in heart muscle cells. Molecular weight of cTnI is 23,875 Dalton consisting of 209 amino acids. [1,2] The cTnI have been used in the diagnosis of acute myocardial infarction(AMI). [3,4,5] According to ESC / ACCF / AHA / WHF, diagnosis of acute myocardial infarction rely on the data from clinical symptoms, Electrocardiogram (EKG) changes in the specific pattern, such as ST-segment elevation / depression, new left bundle branch block, and cardiac biomarker level rise over the 99th percentile upper reference limit, which makes the cTnI level was used to help in making diagnosis for patient coming with symptoms of angina in emergency room.

The current cTnI detecting test has developed more and more high sensitive(called "high-sensitive troponin-I; hsTnI") which can detected in the range 10-50,000 pg / ml (ng / L) [6], and it can detected cTnI level even in normal people unlike cTnI, which only reported positive or negative or lower than the limit of detection. Due to ARCHITECT stat High sensitive Troponin-I (Abbott diagnostic) capabilities, hsTnI level can be detected in normal people up to 96 percent.[7] The reference range of hsTnI which has been researched by Apple FS, et al.(2012) studying the 19 types of cardiac troponin I and T measurement was established. The 99th percentile values for general healthy population without hypertension, diabetes, kidney disease and myocardial infarction, aged 18-64 years was 36 ng / L in men (N = 272), 15 ng / L in women (N = 252) [7].

However, research to find the reference of hsTnI in some groups , especially in patients with kidney disease is still limited and the diagnosis of acute myocardial infarction also use the 99th percentile as the reference source which was researched in healthy population[7] which makes it difficult to interpret. Sometimes doctors may concluded that patients with rising hsTnI because of kidney disease. According to the research in the next section, there are both support and against in this idea. Therefore, the researchers aim to study hsTnI in patients with end-stage renal disease received hemodialysis compare with normal population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more.
* was diagnosed as End-stage renal disease for more than one year.
* Attend hemodialysis 3 times a week consistently for more than 6 months.
* Hemodialysis with Kt/V > 1.2
* No urine output or is less than 500 ml per day.
* No symptoms of myocardial infarction Or were hospitalized with the similar diagnosis during the two weeks.

Exclusion Criteria:

* Could not complete hemodialysis, or Kt / V <1.2
* Has symptoms of myocardial infarction while receiving dialysis
* Has the abnormal symptom (fever, chill, low BP) While receiving dialys

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ESRD group End-stage renal disease patients receiving regular hemodialysis at King Chulalongkorn memorial hospital, Bhumirajanagarindra kidney institute hospital.
  Control group Patients who come to OPD at King Chulalongkorn memorial hospital for their follow up blood check.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
High Sensitive Troponin-I in ESRD group vs Control group | 10 months
  ESRD group
  * Measure the High Sensitive Troponin-I level before the hemodialysis session Control group
  * Measure the High Sensitive Troponin-I as an additional test to their follow up blood check.

SECONDARY OUTCOMES:
High Sensitive Troponin-I in pre-hemodialysis vs post-hemodialysis | 4 hours
  Measure the High Sensitive Troponin-I level before the hemodialysis session comparing to the level after the hemodialysis session.

CONTACTS AND LOCATIONS:
Overall Officials: Khajohn Tiranathanagul, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No